CLINICAL TRIAL: NCT00086359
Title: A Phase III Randomized Trial of the Safety and Antiretroviral Effects of Zidovudine/Lamivudine/Abacavir Versus Zidovudine/Lamivudine/Lopinavir/Ritonavir in the Prevention of Perinatal Transmission of HIV
Brief Title: Comparison of Anti-HIV Drug Combinations to Prevent Mother-to-Child Transmission of HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P1039; 10046 (Registry Identifier: DAIDS ES); PACTG P1039
Record Dates: First submitted 2004-06-30; First posted 2004-07-01 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Perinatal Transmission; Mother-to-Child Transmission; MTCT; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — abacavir; Lamivudine; Zidovudine; lamivudine, zidovudine drug combination; Lopinavir

ARMS (2):
- A (Experimental): One pill of abacavir/lamivudine/zidovudine twice daily
  Interventions: Drug: Abacavir sulfate, lamivudine, and zidovudine
- B (Experimental): One pill of zidovudine/lamivudine and four pills of lopinavir/ritonavir twice daily.
  Interventions: Drug: Lamivudine/zidovudine; Drug: Lopinavir/ritonavir

INTERVENTIONS:
Drug: Abacavir sulfate, lamivudine, and zidovudine — one pill twice daily
  Arms: A
Drug: Lamivudine/zidovudine — one pill twice daily
  Arms: B
Drug: Lopinavir/ritonavir — four pills twice daily
  Arms: B

SUMMARY:
Pregnant women infected with HIV who take anti-HIV medications during pregnancy lower the risk of passing HIV to their infants. This study will compare how well two different combinations of anti-HIV medications control HIV in pregnancy, and whether these combinations of drugs are effective in preventing HIV from being transmitted from a pregnant woman to her baby. The two combinations are abacavir/lamivudine/zidovudine (ABC/3TC/ZDV) and zidovudine/lamivudine (ZDV/3TC) plus lopinavir/ritonavir (LPV/RTV).

DETAILED DESCRIPTION:
Antiretroviral therapy (ART) in pregnancy has dramatically reduced the rates of perinatal HIV transmission. Many pregnant women infected with HIV may not meet the criteria for treatment as set forth by the Department of Health and Human Services' guidelines and would not be started on therapy if they were not pregnant. Pregnant women are prescribed a variety of treatment regimens; the optimum regimen for pregnant women who plan to discontinue therapy after delivery is unknown. An optimum regimen would account for the need for maximum viral suppression, minimal fetal toxicity, and preservation of future therapeutic options for the mother. This study will compare an all nucleoside reverse transcriptase inhibitor (NRTI) regimen of ABC/3TC/ZDV with a standard protease inhibitor (PI) regimen of LPV/RTV and 3TC/ZDV. This study was initially designed for women who plan to take antiretrovirals only while pregnant and do not meet the criteria for treatment initiation if not pregnant. However, pregnant women who have taken ART for 180 days or less or have taken ZDV monotherapy for a total of 8 weeks or less prior to entering this study are eligible for Version 2.0 of this study.

Women in this study will be randomly assigned to one of two groups. Women in Group A will receive one pill ABC/3TC/ZDV twice a day. Women in Group B will receive one pill 3TC/ZDV and 4 pills LPV/RTV twice a day. Women will take their assigned medications until they go into labor. Once in labor, women will be given zidovudine through intravenous (IV) infusion; they will stop taking oral zidovudine but will continue with their other medications. After delivery, all infants will be given zidovudine for six weeks.

Women will have study visits every 2 weeks for the first 8 weeks of treatment, and then every 4 weeks until Week 28. Depending on where a woman is in her pregnancy when she enrolls in the study, she will also have study visits at Weeks 20, 28, and 34 of her pregnancy. At each visit, women will have a medical interview, a physical exam, and an obstetrical exam; blood and urine collection will occur at these visits. Mothers will undergo a fetal ultrasound at Week 20. Adherence, health status, and behavior assessments will occur at selected visits prior to delivery.

After delivery, women will stop taking the study medications but will continue to have study visits at approximately 6, 12, 24, 36, 48, and 52 weeks after delivery. Medical history and a physical exam will occur at all visits for mothers postpartum. Blood collection will occur at every postpartum visit; urine collection will occur 12, 24, and 48 weeks postpartum; health status and behavior assessments will occur at most visits postpartum. Infants will have study visits at 2, 16, and 24 weeks after birth. A medical history, physical exam, and laboratory tests will be conducted at the infant study visits. Women will also be asked to enroll their infants in PACTG 219C, a long-term study that follows infants who are born to HIV infected mothers.

ELIGIBILITY:
Note: The pharmacokinetics testing portion of this study has been discontinued in Version 2.0 of this protocol.

Inclusion Criteria for Mothers:

* HIV infected
* Between the 12th and 30th week of pregnancy
* Intend to continue pregnancy
* Viral load less than 55,000 copies/ml within 30 days of study entry
* CD4 count greater than 350 cells/ml within 30 days of study entry
* Have not previously taken anti-HIV medications (women who have taken 8 weeks or fewer of zidovudine are still eligible) OR have taken anti-HIV medication but have been off treatment for more than 180 days
* Intend to stop taking anti-HIV medications after pregnancy
* Willing to have her infant tested for HIV
* Parent or guardian willing to provide informed consent, if applicable
* Have access to a participating site and are willing to be followed for the duration of the study

Exclusion Criteria for Mothers:

* Chemotherapy for active cancer
* Active opportunistic infection or severe medical condition within 14 days of study entry
* Chronic diarrhea within 1 month of study entry or unresolved acute diarrhea within 7 days of study entry
* Certain abnormal laboratory values
* Diabetes mellitus when not pregnant. Participants who have gestational diabetes are not excluded.
* Current alcohol or other substance abuse that, in the opinion of the investigator, may interfere with the study
* Acute hepatitis within 90 days of study entry
* Major birth defects in infant
* Severe skin disorder (e.g., eczema or psoriasis) requiring systemic treatment
* Require certain medications
* Medical condition that may, in the opinion of the investigator, interfere with the study
* Intend to breastfeed

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Proportion of women in each treatment group with virologic suppression to less than 400 copies/ml at 34th week of pregnancy (or last viral load prior to delivery, if delivery occurs before 34th week of pregnancy) while continuing on assigned therapy | at Week 34 of pregnancy

SECONDARY OUTCOMES:
Primary outcome, evaluating ART naive and ART experienced women | throughout study
HIV-related health status of women at delivery, determined by CD4 counts and plasma HIV-1 viral load in the two treatment groups and in ART naive and ART experienced women | throughout study
study treatment adherence and health status by self report | throughout study
HIV-related health status of women postpartum, determined by CD4 counts and plasma HIV-1 viral load | at Months 3, 6 and 12 postpartum and prior to ART treatment
development of HIV-1 genotypic resistance among women in each treatment group | at delivery, Months 3, 6, and 12 postpartum, and in all cases of treatment failure
incidence of abnormal glucose tolerance, gestational diabetes, and abnormal lactate levels during pregnancy in each treatment group | throughout study
incidence of anemia, hypoglycemia, abnormal liver function studies, prematurity, low birth weight, or perinatal HIV transmission among infants born to women in each treatment group | throughout study
predictive value, sensitivity, and specificity of polymorphisms in HLA-B57, HLA-DR7, and HLA-DQ3 in identifying pregnant women at risk for development of ABC hypersensitivity | throughout study
concentration of T cell receptor rearrangement excision DNA circles | at study entry, delivery and 6 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D. Hull, MD, Study Chair — Department of Reproductive Medicine, Division of Perinatal Medicine, University of California, San Diego School of Medicine
Locations (8):
- United States (7):
  - Usc La Nichd Crs, Los Angeles, California
  - UCSD Mother-Child-Adolescent Program CRS, San Diego, California
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Mt. Sinai Hosp. Med. Ctr. - Chicago, Womens & Childrens HIV Program, Chicago, Illinois
  - Bronx-Lebanon CRS, The Bronx, New York
  - Regional Med. Ctr. at Memphis, Memphis, Tennessee
  - Texas Children's Hosp. CRS, Houston, Texas
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Cooper ER, Charurat M, Mofenson L, Hanson IC, Pitt J, Diaz C, Hayani K, Handelsman E, Smeriglio V, Hoff R, Blattner W; Women and Infants' Transmission Study Group. Combination antiretroviral strategies for the treatment of pregnant HIV-1-infected women and prevention of perinatal HIV-1 transmission. J Acquir Immune Defic Syndr. 2002 Apr 15;29(5):484-94. doi: 10.1097/00126334-200204150-00009. PMID 11981365
- [Background] Scarlatti G. Mother-to-child transmission of HIV-1: advances and controversies of the twentieth centuries. AIDS Rev. 2004 Apr-Jun;6(2):67-78. PMID 15332429
- [Background] Sullivan JL. Prevention of mother-to-child transmission of HIV--what next? J Acquir Immune Defic Syndr. 2003 Sep;34 Suppl 1:S67-72. doi: 10.1097/00126334-200309011-00010. PMID 14562860
- [Background] Thorne C, Newell ML. Mother-to-child transmission of HIV infection and its prevention. Curr HIV Res. 2003 Oct;1(4):447-62. doi: 10.2174/1570162033485140. PMID 15049430
- [Background] Tuomala RE, Shapiro DE, Mofenson LM, Bryson Y, Culnane M, Hughes MD, O'Sullivan MJ, Scott G, Stek AM, Wara D, Bulterys M. Antiretroviral therapy during pregnancy and the risk of an adverse outcome. N Engl J Med. 2002 Jun 13;346(24):1863-70. doi: 10.1056/NEJMoa991159. PMID 12063370